CLINICAL TRIAL: NCT05983952
Title: A Prospective, One-arm and Open Clinical Study to Assess Safety and Efficacy of Anti-CD38 Antibody in the Treatment of Antiphospholipid Syndrome With Secondary Thrombocytopenia
Brief Title: Anti-CD38 Antibody Treating APS With Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023035
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-08

CONDITIONS: Antiphospholipid Syndrome; Thrombocytopenia
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention（Anti-CD38 antibody） (Experimental): 10 enrolled subjects: once a week x 8 doses
  Interventions: Drug: Anti-CD38 antibody Injection

INTERVENTIONS:
Drug: Anti-CD38 antibody Injection — intravenous Anti-CD38 antibody administration
  This study adopts a prospective, single arm, open design method. Ten subjects were enrolled in the study and were treated with Anti-CD38 antibody (16mg/kg/w) for 8 weeks.
  The first stage is the main research stage (d1-w8), which is the core treatment period. The subjects will receive intravenous infusion of 16mg/kg Anti-CD38 antibody once a week for 8 weeks to observe the safety and efficacy during treatment.
  The second stage (w9-w24) is the stage of withdrawal from the visit, mainly to observe the safety and continuous efficacy of Anti-CD38 antibody after treatment.

SUMMARY:
To evaluate the safety and efficacy of anti-CD38 antibody in the treatment of antiphospholipid syndrome with secondary thrombocytopenia in patients who have not responded adequately or relapsed after first-line treatment and at least one second-line therapy including rituximab and/or TPO-RA.

DETAILED DESCRIPTION:
The anti-phospholipid syndrome (APS) is a systemic autoimmune disorder characterized by recurrent thrombosis and/or obstetrical morbidity along with persistent anti-phospholipid antibodies (APLA), including lupus anticoagulant (LA), anti-β2-glycoprotein I (anti-β2GPI) and/or anti-cardiolipin (aCL) antibodies. APS is one of the most common acquired thrombophilias, and unlike most of the genetic thrombophilias, ise associated with both venous and arterial thrombosis. The deep veins of the lower extremities and the cerebral arterial circulation are the most commonly affected venous and arterial sites, respectively. It has been posited that "two hits" are necessary to trigger a thrombotic event in antiphospholipid syndrome. This hypothesis argues that antiphospholipid antibodies provide the first hit by creating a generalized procoagulant state, which conspires with a second hit (often cryptic and potentially the result of subclinical vascular injury, stasis, or inflammation) that triggers thrombosis. The evidence that IgG antibodies targeting domain I of β2GPI contribute to the prothrombotic state of antiphospholipid syndrome is convincing. Meanwhile, data also support roles for other isotypes of aβ2GPI, antibodies that target heterotypic complexes of phospholipids and phospholipid binding proteins, and antibodies that target phospholipids directly. Given that most mechanistic studies have focused on either polyclonal IgG fractions isolated from patients with antiphospholipid syndrome or IgG anti-β2GPI, researchers unfortunately could not build a nuanced model of how diverse species of antiphospholipid antibodies conspire to cause various manifestations of antiphospholipid syndrome.

The Sapporo classification criteria for APS were first proposed in 1999, and updated at the Eleventh International Congress on Antiphospholipid Antibodies in Sydney in 2006.Patient must have both clinical and laboratory criteria to meet a diagnosis of APS. Clinical criteria include either objectively confirmed venous, arterial or small vessel thrombosis, or obstetric morbidity including the unexplained death of one or more morphologically normal fetuses at or beyond the 10th week of gestation, the premature birth of one or more morphologically normal neonates before the 34th week of gestation, and/or three or more unexplained, consecutive spontaneous abortions before the 10th week of gestation. Since these clinical manifestations are prevalent in the general population and may have a multifactorial etiology, laboratory investigations are central to the diagnosis of APS. The updated Sydney classification scheme also requires specific laboratory criteria: a lupus anticoagulant detected according to guidelines published by the International Society on Thrombosis and Hemostasis (ISTH), anticardiolipin (aCL) antibodies (IgG or IgM) exceeding 40 IgG or IgM antiphospholipid units, or anti-β2GPI antibodies (IgG or IgM) at levels exceeding the 99th percentile, measured by enzyme-linked immunosorbent assay (ELISA). To minimize the risk of making a diagnosis based on transient ntiphospholipid antibodies, the recommendations are to perform assays on two separate occasions, at least twelve weeks apart.The major changes made in the 2006 revision of the Sapporo criteria were that anti-β2GPI antibody was included for the first time and a recommendation was made to classify patients into those with only one positive APLA and those with two or three positive APLA, based on accumulating information suggesting that positivity in more than a single assay was associated with higher thrombotic risk.

Thrombocytopenia occurs in APS with a frequency ranging from 20% to 50%, and the estimated bleeding risk associated with it is much lower than the thrombotic risk associated with aPL. In some patients with a confirmed APS diagnosis, secondary immune thrombocytopenia (ITP) may lead to severe thrombocytopenia with consequent major bleeding. At the same time, the presence of antiphospholipid antibodies (aPL) in patients with a diagnosis of primary ITP has been reported in several studies, although with some specific characteristics especially related to the variety of antigenic targets. Even though it does not enter the APS defining criteria, thrombocytopenia should be regarded as a warning sign of a "high risk" APS and thus thoroughly evaluated. The presence of aPL in patients with ITP should be assessed as well to stratify the risk of paradoxical thrombosis. In detail, besides the high hemorrhagic risk in secondary thrombocytopenia, patients with a co-diagnosis of APS or only antibodies are also at risk of arterial and venous thrombosis. The pathogenesis of thrombocytopenia in antiphospholipid antibody-positive patients is not fully understood. However, based on currently available data, four different pathogenesis hypothesis were proposed, including secondary Immune thrombocytopenia, decreased platelet production, increased platelet pooling and increased platelet consumption. The APS associated thrombocytopenia treatment guidelines can be drawn lessons from the treatment strategies of ITP. Conventional treatment of adult APS associated thrombocytopenia includes first-line glucocorticoid and immunoglobulin therapy. B-cell targeted drugs are effective in the treatment of APS. Studies have found that rituximab can improve the clinical manifestations (including thrombocytopenia) and serological indicators in the late stage of APS treatment. Splenectomy is reserved for refractory patients who present with severe bleeding symptoms and are resistant to glucocorticoids and immunosuppressants. Plasmapheresis can be used in patients with CAPS when severe thrombocytopenia occurs. Thrombopoietin receptor agonists may increase the risk of thrombosis in APS patients and should be used with caution. When thrombosis coexists with bleeding events associated with thrombocytopenia, if platelet counts reach safe levels (> 50×109/L), glucocorticoid combined with anticoagulant therapy is recommended. It is difficult to treat APS patients with severe thrombocytopenia and severe bleeding. It has been reported in previous literature that platelets can be significantly increased in some patients after treatment with hormones or rituximab, immunosuppressants, etc., but it is easy to relapse and difficult to maintain. The decrease of aPL is not obvious and it is difficult to completely remove. It is a difficult point in the treatment of hematology.

Anti-CD38 antibody, which targets plasma cells, has been used in multiple myeloma in a number of clinical studies and has shown good therapeutic effects. In addition, the clinical trials of anti-CD38 antibody analogues such as fizumatumumab in the treatment of autoimmune diseases including membranous nephropathy and systemic lupus erythematosus (SLE) are also being carried out simultaneously. A case report of anti-CD38 antibody in the treatment of APS has been reported abroad, and it has been found that it can significantly reduce the titer of antiphospholipid antibodies. In the process of treating ITP patients with antiphospholipid antibodies, investigators found that anti-CD38 antibody could not only rapidly increase platelet count, but also significantly reduce the titer of antiphospholipid antibodies, which may have a significant therapeutic effect on APS.Therefore, the use of daratumumab to clear APS with secondary thrombocytopenia may be effective and represents a new therapeutic strategy.

Therefore, the investigators designed this clinical trial to evaluate the safety and efficacy of anti-CD38 antibody in the treatment of antiphospholipid syndrome with secondary thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female.
* Conform to the diagnostic criteria of antiphospholipid syndrome (APS).
* Failure to achieve response or relapse after corticosteroid therapy, and at least one second-line therapy including rituximab, CSA or CTX etc., or those who cannot chose other second-line therapy.
* Platelet count of <30 X 10^9/L.
* With normal hepatic and renal functions.
* ECOG physical state score ≤ 2 points.
* Cardiac function of the New York Society of Cardiac Function ≤ 2.
* Signed and dated written informed consent

Exclusion Criteria:

* Received any treatment of anti-CD38 antibody drug
* Uncontrollable primary diseases of important organs, such as malignant tumors, liver failure, heart failure, renal failure and other diseases;
* HIV positive;
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C, cytomegalovirus, EB virus and syphilis positive;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc.;
* At present, there are heart diseases, arrhythmias that need treatment or hypertension that researchers judge is poorly controlled;
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis and atherosclerosis;
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past;
* Patients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up;
* Patients whose toxic symptoms caused by pre-trial treatment have not disappeared;
* Other serious diseases that may limit the subject's participation in this test (such as diabetes; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer, etc.);
* Patients with septicemia or other irregular severe bleeding;
* Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy after anti-CD38 antibody treatment within 8 weeks | 8 weeks
  Proportion of subjects with a platelet count ≥ 50 × 10^9/L within 8 weeks after initial administration in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period
Safety of anti-CD38 antibody | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after anti-CD38 antibody treatment

SECONDARY OUTCOMES:
Response rate of treatment | 12 weeks
  Including: 1. Proportion of subjects with a platelet count ≥ 50 × 10^9/L at week 2, week 4, week 6，week 8，week 10 and week 12 in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the study period; 2. Proportion of subjects achieving platelet counts ≥ 50×10^9/L at least once in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids during the first 12 weeks; 3. Proportion of subjects whose platelet counts ≥ 30×10^9/L and at least two times of baseline platelet count in absence of rescue therapy, and without having had dose increment of TPO-RA or corticosteroids within 8 weeks（two consecutive measurements at least 7 days apart）.
Duration from treatment initiation to platelet count ≥50×10^9/L | 12 weeks
  Duration from treatment initiation to platelet count ≥50×10^9/L without having received any platelet elevating therapy or having had dose increment of TPO-RA and/or corticosteroids
Duration of platelet response | 24 weeks
  The longest duration for which the subject sustained a platelet count ≥50×109/L
platelet count ≥50×10^9/L ≥75% tests | 24 weeks
  Proportion of subjects with platelet count ≥50×10^9/L in ≥ 75% of the total number of tests
Measurements of platelet count at each visit time point | 24 weeks
  Platelet count at each visit time point
Emergency treatment | 24 weeks
  Percentage of subjects who received emergency treatment
Number of subjects with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | 24 weeks
  Changes of the subjects' numbers in WHO bleeding score after Anti-CD38 antibody treatment according to the reported World Health Organization's Bleeding Scale. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Occurrence of thrombosis | 24 weeks
  Assessment of the occurrence of thrombosis during the study period
Measurements of antiphospholipid antibody | 24 weeks
  Measurements of the level of antiphospholipid antibody during the study period
platelet count ≥50×10^9/L at least once | 8 weeks
  Percentage of subjects with a platelet count ≥50×109/L at least once 8 weeks after the first dose
platelet count ≥30×10^9/L and at least 2-fold from baseline on at least one occasion | 8 weeks
  The percentage of subjects with a platelet count ≥30×10^9/L and at least 2-fold from baseline 8 weeks after the first dose on at least one occasion
Measurements of various subsets of immunocompetent cells | 24 weeks
  To assess the changes of the percentage of B cell subsets，regulatory B cells（Breg），regulatory T cells (Treg)，supressor T cells（Ts），monocyte subcets, helper T cells（Th）subsets and the functionally-polarized CD4+ T cell subsets, etc. in peripheral blood mononuclear cells（PBMCs）before and after anti-CD38 antibody therapy, and to compare with the healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI